CLINICAL TRIAL: NCT02516449
Title: Utility of Two Patients Decision Aids About Asthma Inhaled Controller Medication Use in Adult Patients With Asthma
Brief Title: Assessment of Shared Decision Making Aids in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Chaire en transfert de connaissances, éducation et prévention en santé respiratoire et cardiovasculaire de l'Université Laval (Unknown); Chaire sur l'adhésion aux traitements de l'Université Laval (Unknown); Chaire de recherche du Canada en implantation de la prise de décision partagée dans les soins primaires de l'Université Laval (Unknown)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD FRCPC FCCP, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CER 20858
Record Dates: First submitted 2015-07-02; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient decision aids (Experimental): Participants read and fill a patient decision aid before being provided education on asthma.
  Interventions: Other: Patient decision aid
- Usual care (No Intervention): Participants do not read and fill a patient decision aid before being provided education on asthma.

INTERVENTIONS:
Other: Patient decision aid — The patient decision aid is a 12-page A3 size color-printed booklet entitled "Should I take asthma inhaled controller medication to optimize asthma control?"
  Arms: Patient decision aids

SUMMARY:
The purpose of this study is to determine whether the use of shared decision making aids is more effective than usual care in improving asthma knowledge, lessening decisional conflict, and enhancing adherence to treatments and asthma control in adult patients with mild to severe asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, aged 18 to 65 years;
2. Current diagnosis of mild to severe asthma; 2.1) Asthma diagnosis will be made upon one of the following criteria: 2.1.1) Forced expiratory volume in one second (FEV1) increases by at least 12% after the use of a bronchodilator (and a minimum ≥ 200 mL); 2.1.2) Current asthma symptoms and a positive methacholine challenge test (20% fall in FEV1 after inhalation of a provocative dose of methacholine 16 mg/mL); 2.1.3) A respirologist's current diagnosis of asthma found in the patient's medical report. 2.2) Severity of asthma will be assessed according to prescribed pharmacotherapy, as suggested by the 2012 Canadian Thoracic Society Guidelines: 2.2.1) Patients with mild asthma using SABA as well as low doses (≤250 mcg/day beclomethasone or equivalent) of inhaled glucocorticosteroids; 2.2.2) Patients with moderate asthma using SABA as well as low to moderate doses (250mcg/day < dose ≤500 mcg/day beclomethasone or equivalent) of inhaled glucocorticosteroids, with or without additional therapy (LABA or LTRA); 2.2.3) Patients with severe asthma using high doses (>500 mcg/day beclomethasone or equivalent) of inhaled glucocorticosteroids, and additional pharmacotherapy (LABA, LTRA, or Prednisone), and SABA.

Exclusion Criteria:

1. Chronic obstructive pulmonary disease (COPD);
2. Education on asthma in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in asthma knowledge at 2 months, measured by QCALF score | Visit 1 (baseline) and visit 2 (2-month follow-up)
Change from baseline in decisional conflict at 2 months, measured by DCS score | Visit 1 (baseline) and visit 2 (2-month follow-up)

SECONDARY OUTCOMES:
Change from baseline in adherence to treatment at 2 months, measured by questionnaire | Visit 1 (baseline) and visit 2 (2-month follow-up)
Change from baseline in asthma control at 2 months, measured by ACSS score | Visit 1 (baseline) and visit 2 (2-month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada